CLINICAL TRIAL: NCT04858685
Title: Determination of Factors Affecting Early Mobilization of Patients Who Have Undergone Knee and Hip Arthroplasty
Brief Title: Early Mobilization After Arthroplasty
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, AKİF BULUT, Principal Investigator, Uludag University
Other Study IDs: 2017-14/26
Record Dates: First submitted 2021-04-07; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Mobility
Keywords: Early Mobilization; Enhanced Recovery After Surgery (ERAS); Arthroplasty; Nursing
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: early mobilization — early mobilization was defined, on the basis of the ERAS protocol, as mobilization of a few steps or a few meters from the bed within the first 24 hours after surgery with another person's support/control and/or a walking aid.

SUMMARY:
Aims and Objectives: This study was conducted in order to determine the factors that affected the early mobilization after surgery of patients who had undergone knee and hip arthroplasty.

Background: Early mobilization in knee and hip arthroplasty is still not at the desired level, and it is among the most frequently overlooked nursing practices.

Desing: This study is descriptive and cross-sectional. STROBE checlist was used to compile the study's report.

Methods: The universe of the study consisted of a total of 80 patients who were hospitalized between 07 November 2017 and 21 September 2018 in the Orthopedics and Traumatology Clinic of a State Hospital to undergo knee or hip arthroplasty, and who met the inclusion criteria. The sample of the study consisted of 60 patients who were in the universe of the study, who met the inclusion criteria and who voluntarily agreed to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Orthopedics and Traumatology Clinic for the first time to undergo knee or hip arthroplasty,
* Communicating,
* No hearing or speech impairment,
* 18 years and older patients.

Exclusion Criteria:

* Undergoing revision surgery,
* Having a history of lower extremity orthopedic intervention that may prevent mobilization,
* Having neurological and medical problems that may cause locomotor disability,
* Uncontrollable heart and lung diseases,
* Having a history of neurological disease (Alzheimer's, dementia, etc.),
* Patients with gout, metabolic diseases or septic arthritis.

Ages: 48 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The universe of the study consisted of a total of 80 patients who were hospitalized between November 2017 and September 2018 in the Orthopedics and Traumatology Clinic of a State Hospital to undergo knee or hip arthroplasty, and who met the inclusion criteria. The improbable sampling method was used in the study. The sample of the study consisted of 60 patients who were in the universe of the study, who met the inclusion criteria and who voluntarily agreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The status of successful mobilization within 24 hours after surgery | 24 Hours
  Early mobilization was defined, on the basis of the ERAS protocol, as mobilization of a few steps or a few meters from the bed within the first 24 hours after surgery with another person's support/control and/or a walking aid.

CONTACTS AND LOCATIONS:
Overall Officials: AKİF BULUT, Phd Student, Principal Investigator — Uludag University
Locations (1):
- Karacabey State Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to carry out the study, it has been determined that the data will not be shared with anyone else with the permission of the provincial health directorate.

REFERENCES:
- [Derived] Bulut A, Vatansever NA. Determination of Factors Affecting Early Mobilization of Patients Who Have Undergone Knee and Hip Arthroplasty. J Perianesth Nurs. 2022 Oct;37(5):646-653. doi: 10.1016/j.jopan.2021.10.013. Epub 2022 May 4. PMID 35525826

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT04858685/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT04858685/ICF_001.pdf